CLINICAL TRIAL: NCT01549613
Title: Evaluation of Daptomycin for the Emergency Department Treatment of Complicated Skin and Skin Structure Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, George Shaw, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-11-03-06
Record Dates: First submitted 2012-02-08; First posted 2012-03-09 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Cellulitis; Skin Infections
MeSH Terms: conditions — Cellulitis | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard treatment with daptomycin (Active Comparator): Daptomycin will be given in a one-time dose of 4mg/kg in a one-time dose to be infused over 2 minutes at the initiation of patient therapy in the RDTC cellulitis protocol
  Interventions: Drug: Daptomycin
- standard treatment of vancomycin (Active Comparator): Vancomycin will be given in a dose of 15mg/kg at baseline and again at 12 hours to be infused over 1 to 2 hours.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Daptomycin — • Daptomycin will be given in a one-time dose of 4mg/kg in a one-time dose to be infused over 2 minutes at the initiation of patient therapy in the RDTC cellulitis protocol.
  Arms: standard treatment with daptomycin
Drug: Vancomycin — • Vancomycin will be given in a dose of 15mg/kg at baseline and again at 12 hours to be infused over 1 to 2 hours.
  Arms: standard treatment of vancomycin

SUMMARY:
This is a prospective, randomized clinical trial comparing daptomycin to vancomycin in the Emergency Department (ED) treatment of complicated skin and skin structure infection in the Rapid Diagnosis and Treatment Center (RDTC). In brief, a convenience sample of patients who are admitted to the RDTC cellulitis protocol in the ED will be randomized to either vancomycin, which is currently an accepted care standard in the RDTC cellulitis protocol, or daptomycin, which is the experimental treatment in this study. The primary hypothesis is that daptomycin treatment is as efficacious as standard therapy in the treatment of ED cellulitis.

DETAILED DESCRIPTION:
Specific Aim 1: Compare the efficacy of daptomycin to the efficacy of vancomycin for the treatment of complicated skin and skin structure infection in the ED. Patients eligible for the RDTC Cellulitis Treatment Protocol will be screened for inclusion in the study. After informed consent, patients will be randomized to receive either daptomycin or vancomycin (1:1 ratio). A case report form (CRF) detailing medical history, clinical characteristics, and treatments will be completed. The patients will be evaluated for meeting RDTC discharge criteria. The following time points will be collected: 1. actual time patient meets discharge criteria based on the RDTC cellulitis protocol; 2. time of disposition defined as the time treating physician writes discharge orders; and, 3. time the patient actually leaves the emergency department. Subsequently, the patient will be followed up by telephone to ascertain whether a change in antibiotic therapy or a return ED visit for complicated skin and skin structure infection occurred within 30 days of the initial RDTC enrollment Specific Aim 2: Compare the change in area and erythema of the cellulitic lesion between patients treated with daptomycin and patients treated with vancomycin. Patients enrolled in the study will have serial digital photographs of their primary lesion taken. The images will be processed blinded to clinical data and asynchronous to the ED stay. The change in lesion area and erythema will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to RDTC to the Cellulitis Protocol
* 18 yrs old or greater
* Able and willing to give informed consent
* Hemodynamically stable (systolic blood pressure >90mmHg and heart rate <120 beats per minute)

Exclusion Criteria:

* Antibiotics given prior to enrollment
* Suspected necrotizing infection
* Diabetic foot ulcer
* Genitourinary involvement
* Post operative infection (not including simple wound closure infection)
* Suspected gouty or septic arthritis
* Chronic Lymphangitis
* Requiring routine hemodialysis
* Patient reported allergy to Vancomycin
* Patient reported allergy to Daptomycin
* Participation in another investigational treatment study within 30 days prior to enrollment
* Prisoner
* Pregnant or breast-feeding
* Complicated skin and skin structure infection of the face

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George J. Shaw, MD, PhD, Principal Investigator — University of Cincinnati, Dept. of Emergency Medicine
Locations (1):
- University of Cincinnati, Dept. of Emergency Medicine, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Treatment With Daptomycin | Standard Treatment of Vancomycin
Started | 50 | 50
Completed | 39 | 39
Not Completed | 11 | 11
Not completed — Lost to Follow-up | 11 | 11

BASELINE CHARACTERISTICS:
Population: 161 patients were screened;104 were initially enrolled. 3 patients were withdrawn prior to randomization; 1 patient was transferred to OR, 1 patient was admitted prior to randomization, 1 patient was prescribed a different antibiotic;1 patient was withdrawn not meet inclusion criteria. 39 patients in each treatment group completed follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment With Daptomycin | Standard Treatment of Vancomycin | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 38 (13) | 40 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 29 | 35 | 64
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 14 | 34
  White | 29 | 34 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction of Discharge Criteria
Description: RDTC cellulitis protocol discharge criteria
Time Frame: Time point at which outcome measure is assessed 30 days from the date of admission.
Measure: Number; unit: participants
Arm/Group | Standard Treatment With Daptomycin | Standard Treatment of Vancomycin
Number analyzed (Participants) | 50 | 50
participants | 15 [-0.58 to 1.98] | 14

2. Secondary Outcome: Digital and Infrared Imaging
Description: Change in lesion area and temperature
Time Frame: Time frame begins on admission to RDTC for cellulitis and measurements will be taken every 2hour times 2 and every 4 hours until discharge from the RDTC.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Standard Treatment With Daptomycin | Standard Treatment of Vancomycin
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 4/50 | 7/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment With Daptomycin (N=50) | Standard Treatment of Vancomycin (N=50)
hospital readmission (Investigations) | 1 (1) | 2 (2) — returned to hospital within 30 days
redman syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Developed reaction to antibiotic
Sought treatment of town (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Patient reported that they went to doctor in home town for further treatment
hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — developed hives during course of treatment
scheduled surgery for ovarian cyst (General disorders) | 1 (1) | 0 (0) — The surgery date was moved a week later after completing antibiotic
Returned to pmc for HPT and Diabetes (General disorders) | 1 (1) | 0 (0) — Patient admitted to medical service for hyperkalemia
Iv infiltrated (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — IV infiltrated while antibiotic infusing.
dog bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — patient obtain dog bite after enrollment and returned to ED for treatment
Red streak (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — a red streak from cellulitis to arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No